CLINICAL TRIAL: NCT00508820
Title: An Open Label Study of Romiplostim in Adult Thrombocytopenic Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Brief Title: An Open Label Study of Romiplostim in Adult Thrombocytopenic Subjects With ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040209
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Thrombocytopenia; Thrombocytopenic Purpura
Keywords: Platelet; AMG 531; Thrombopoietin; blood disorder; bleeding disorder; immune thrombocytopenic purpura; idiopathic thrombocytopenic purpura; immune (idiopathic) thrombocytopenic purpura; TPO; thrombopoietic protein
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Purpura, Thrombocytopenic; Jacobs syndrome; Hematologic Diseases; Hemostatic Disorders | interventions — romiplostim

ARMS (1):
- 1 (Experimental): Romiplostim
  Interventions: Biological: Romiplostim

INTERVENTIONS:
Biological: Romiplostim — Romiplostim will be administered subcutaneously QW. Romiplostim will be manufactured and packaged and distributed using Amgen's clinical study investigational product distribution procedures. Romiplostim is presented as a lyophilized, white powder in 5.0 mL glass vials.

SUMMARY:
This protocol will provide open label romiplostim to adult thrombocytopenic subjects. Romiplostim will be administered by subcutaneous injection once per week. Dose adjustment will be based on platelet counts, and will be allowed throughout the duration of the study. Rescue therapies are allowed at any time during the study. Reductions in concurrent ITP therapies may occur at any time when platelet counts are > 50,000.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject has a diagnosis of immune (idiopathic) thrombocytopenic purpura per the American Society of Hematology guidelines
* If Subject is > 60 years of age, subject has a written bone marrow aspiration and/or biopsy report consistent with a diagnosis of ITP
* Subject has received at least 1 prior therapy for ITP
* Subject's platelet count is ≤ 30,000 or the subject is experiencing bleeding that is uncontrolled with conventional therapies
* Subject (or legally-acceptable representative) is willing and able to provide written informed consent

Exclusion Criteria:

* Subject has a history of hematological malignancy, myeloproliferative disorder, myelodysplastic syndrome (MDS), or bone marrow stem cell disorder
* Subject has participated in any study evaluating PEG-rHuMGDF, recombinant human thrombopoietin (rHuTPO), or related platelet product
* Subject has a known hypersensitivity to any recombinant E coli-derived product
* Subject has received any therapeutic drug or device that is not approved by the local regulatory health agency for any indication within 4 weeks of Screening
* Subject is of reproductive potential and is not using adequate contraceptive precautions, in the judgment of the investigator
* Subject is pregnant or breast feeding
* Investigator has concerns regarding the subject's ability to comply with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Janssens A, Tarantino M, Bird RJ, Mazzucconi MG, Boccia RV, Fernandez MF, Kozak T, Steurer M, Boekhorst Pt, Dillingham K, Kreuzbauer G, Woodard P. Romiplostim Treatment in Adults with Immune Thrombocytopenia of Varying Duration and Severity. Acta Haematol. 2015;134(4):215-28. doi: 10.1159/000381657. PMID 26066765
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 24Feb2005 Last Subject Enrolled: 05Jan2010
Groups:
- Romiplostim (AMG 531) Cohort 1: Romiplostim administered to participants subcutaneously weekly based on platelet counts. Participants were enrolled under the original protocol or protocol amendments 1-3 where starting dose was 3mcg/kg.
- Romiplostim (AMG 531) Cohort 2: Romiplostim administered to participants subcutaneously weekly based on platelet counts. Participants were enrolled under protocol amendments 4 where starting dose was 1mcg/kg.
Period: Overall Study
Arm/Group | Romiplostim (AMG 531) Cohort 1 | Romiplostim (AMG 531) Cohort 2
Started | 168 | 239
Completed | 113 | 175
Not Completed | 55 | 64
Not completed — Adverse Event | 6 | 10
Not completed — Death | 6 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 8 | 2
Not completed — Pregnancy | 0 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Other | 11 | 2
Not completed — Noncompliance | 1 | 0
Not completed — Requirement for alternative therapy | 7 | 15
Not completed — Protocol-specified Criteria | 3 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Romiplostim (AMG 531) Cohort 1 | Romiplostim (AMG 531) Cohort 2 | Total
Number analyzed (Participants) | 168 | 239 | 407
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (17) | 54.1 (18) | 53.9 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 150 | 244
  Male | 74 | 89 | 163
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 149 | 232 | 381
  Black or African American | 5 | 1 | 6
  Hispanic or Latino | 7 | 2 | 9
  Asian | 5 | 3 | 8
  Other | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: One or more occurences of one or more adverse events within the participant during the study. Participants with more than one event were only counted once
Time Frame: Duration of Treatment plus 30 days or End of Study (whichever is later). Approximately 205 weeks.
Population: Safety Analysis Set, comprised of all participants who received at least one dose of romiplostim
Measure: Number; unit: participants
Arm/Group | Romiplostim (AMG 531) Cohort 1 | Romiplostim (AMG 531) Cohort 2
Number analyzed (Participants) | 168 | 239
participants | 162 | 215

2. Secondary Outcome: Platelet Response (Definition 1)
Description: Platelet response using definition1 . (a doubling of baseline platelet count and a platelet count of >=50 x 10^9/L
Time Frame: Duration of treatment (up to 201 weeks)
Population: Full Analysis Set, all enrolled participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim (AMG 531) Cohort 1 | Romiplostim (AMG 531) Cohort 2
Number analyzed (Participants) | 168 | 239
Participants | 156 | 214

3. Secondary Outcome: Platelet Response (Definition 2)
Description: Platelet response using definition 2 (a platelet count increase of >=20 x 109/L from baseline)
Time Frame: Duration of treatment (up to 201 weeks)
Population: Full Analysis Set, all enrolled participants
Measure: Number; unit: Participants
Arm/Group | Romiplostim (AMG 531) Cohort 1 | Romiplostim (AMG 531) Cohort 2
Number analyzed (Participants) | 168 | 239
Participants | 160 | 220

ADVERSE EVENTS:
Time Frame: Average duration: cohort 1 52 wks; cohort 2 42 wks.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Romiplostim Cohort 1 | Romiplostim Cohort 2
Serious Adverse Events (participants affected / at risk) | 61/168 | 61/239
Other Adverse Events (participants affected / at risk) | 155/168 | 188/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim Cohort 1 (N=168) | Romiplostim Cohort 2 (N=239)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow disorder (Blood and lymphatic system disorders) | 0 | 1
Bone marrow reticulin fibrosis (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 5 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 10
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Hyperpyrexia (General disorders) | 0 | 1
No therapeutic response (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Sudden death (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 2
Acute tonsillitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 3
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood smear test abnormal (Investigations) | 0 | 1
Electrocardiogram (Investigations) | 1 | 0
Platelet count abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 2
Troponin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Dementia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Mononeuropathy multiplex (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Temporal lobe epilepsy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 2
Purpura (Skin and subcutaneous tissue disorders) | 3 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim Cohort 1 (N=168) | Romiplostim Cohort 2 (N=239)
Anaemia (Blood and lymphatic system disorders) | 13 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 11
Abdominal pain (Gastrointestinal disorders) | 18 | 11
Constipation (Gastrointestinal disorders) | 20 | 12
Diarrhoea (Gastrointestinal disorders) | 33 | 24
Dyspepsia (Gastrointestinal disorders) | 9 | 5
Gingival bleeding (Gastrointestinal disorders) | 14 | 5
Mouth haemorrhage (Gastrointestinal disorders) | 11 | 15
Nausea (Gastrointestinal disorders) | 32 | 38
Vomiting (Gastrointestinal disorders) | 12 | 11
Asthenia (General disorders) | 13 | 18
Chest pain (General disorders) | 10 | 7
Chills (General disorders) | 11 | 4
Fatigue (General disorders) | 50 | 25
Influenza like illness (General disorders) | 11 | 8
Oedema peripheral (General disorders) | 24 | 23
Pain (General disorders) | 16 | 7
Pyrexia (General disorders) | 19 | 13
Influenza (Infections and infestations) | 9 | 25
Nasopharyngitis (Infections and infestations) | 38 | 31
Rhinitis (Infections and infestations) | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 24 | 14
Urinary tract infection (Infections and infestations) | 11 | 8
Viral infection (Infections and infestations) | 15 | 1
Contusion (Injury, poisoning and procedural complications) | 39 | 21
Decreased appetite (Metabolism and nutrition disorders) | 16 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 28
Dizziness (Nervous system disorders) | 28 | 15
Headache (Nervous system disorders) | 57 | 61
Hypoaesthesia (Nervous system disorders) | 9 | 0
Paraesthesia (Nervous system disorders) | 10 | 16
Anxiety (Psychiatric disorders) | 11 | 5
Depression (Psychiatric disorders) | 10 | 7
Insomnia (Psychiatric disorders) | 19 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 14
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 29 | 31
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 12
Rash (Skin and subcutaneous tissue disorders) | 17 | 8
Haematoma (Vascular disorders) | 8 | 17
Hypertension (Vascular disorders) | 13 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.